CLINICAL TRIAL: NCT01562782
Title: Fructose-induced Hepatic De Novo Lipogenesis in South Asians
Brief Title: Change of Fructose to Fat in South Asians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1110011995
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Elevated Triglycerides; Diabetes; Cardiovascular Disease; Dyslipidemia
Keywords: Elevated triglycerides; Diabetes Mellitus; Dyslipidemia; Lipid Metabolic Disorders; Body Weight
MeSH Terms: conditions — Hypertriglyceridemia; Diabetes Mellitus; Cardiovascular Diseases; Dyslipidemias; Body Weight | interventions — Fructose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- South Asians (Experimental): Participants in this group have only South Asian heritage. The intervention is Fructose + Glucose Beverage.
  Interventions: Other: Fructose + Glucose Beverage
- Caucasians (Active Comparator): Participants in this group have only Caucasian heritage. The intervention is Fructose + Glucose Beverage.
  Interventions: Other: Fructose + Glucose Beverage

INTERVENTIONS:
Other: Fructose + Glucose Beverage — Consumption of a sweet beverage (Fructose:Glucose 1:1, 3g/kg) over 1/2 hour. Blood sampling will occur before and after consumption of beverage.

SUMMARY:
The purpose of this study is to determine whether hepatic de novo lipogenesis (DNL) in response to the ingestion of a mixture of glucose and fructose is greater in South Asians compared to controls (Caucasians).

DETAILED DESCRIPTION:
South Asians, who originate from the Indian subcontinent and make up one-fifth of the world's population, are among the highest number who suffer from heart disease and diabetes. The results of many research studies suggest that genes play a role in developing heart disease and diabetes that is made worse by the diet in the United States. Fructose is a sugar widely used in the American diet, and when consumed, it is taken up by the liver and changed into fats through a process called de novo lipogenesis (DNL). The current study will compare this change into fats in the liver between South Asians and Caucasians. The participants will be screened on the initial visit, and on the second visit, the DNL response will be measured in the blood over four hours after drinking one sweetened beverage, containing half glucose, half fructose, similar to a soft drink. We expect that DNL in response to fructose intake is higher in South Asians when compared to Caucasians and may partially explain why South Asians have earlier heart disease and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-35 years of age.
* South Asian or Caucasian descent through self-identification (South Asians are to have both biological parents with ancestry from India, Pakistan, Sri Lanka, Nepal and Bangladesh and no known non-South Asian ancestry in parents; Caucasians are to have both biological parents who self-identify as Caucasian and no known non-Caucasian ancestry in parents).
* Body mass index (BMI) 18.0-24.9 kg/m2 with no history of obesity.
* Fasting glucose <100 mg/dL, 2h glucose oral glucose tolerance test (OGTT) < 140 mg/dL.
* triglycerides (TG) <200 mg/dL, HDL cholesterol (HDL-C) >30 mg/dL, LDL cholesterol (LDL-C) <160 mg/dL.
* Willing and able to stop fish oil, fiber supplement, other non-prescribed vitamins/supplements for 1 week prior to visit #2 until completion of study.
* Willing to not drink alcohol for 24-hours before visit #2.
* Willing and able to provide informed consent.

Exclusion Criteria:

* History of diabetes or other endocrine disorder, hepatitis or other liver disorder, HIV, or autoimmune disease.
* Medication(s) known to affect lipids, including hormonal contraceptives.
* Recent acute illness
* Gastrointestinal disease resulting in significant gastrointestinal dysfunction or malabsorption.
* Cigarette smoking
* History of ethanol abuse (current intake >2 drinks/day) or illicit drugs.
* History of severe psychiatric illness
* If female, pregnant or breastfeeding
* Participation in an investigational drug study within one month of screening.
* Unusual diet or extreme level of physical activity
* Have any other condition, which in the opinion of the investigator, should prohibit the participation in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-04-02 (Actual); Primary Completion 2013-10-10 (Actual); Study Completion 2013-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hudgins, MD, Principal Investigator — The Rogosin Institute
Locations (2):
- United States (2):
  - The Rogosin Institute, New York, New York
  - Weill Cornell Medical College Clinical and Translational Science Center (CTSC), New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 4/2012 and 10/2013 fifteen South Asians and 15 Caucasians were studied as outpatients at the Weill Cornell Medical College Clinical and Translational Science Center (CTSC).
Pre-assignment Details: At the CTSC clinic, consented volunteers had their medical history reviewed and a physical exam performed. A fasting blood sample was obtained to screen for lipid and biochemical abnormalities, thyroid and liver disease, anemia, pregnancy and diabetes/glucose intolerance.
Groups:
- Caucasians: Control group: The arm is an oral sugar challenge with blood sampling over 4 hours.
  Fructose + Glucose Beverage: Consumption of a sweet beverage (Fructose:Glucose 1:1, 3g/kg) over 1/2 hour. Blood sampling will occur before and after consumption of beverage.
- South Asians: South Asian group: The arm is an oral sugar challenge with blood sampling over 4 hours.
  Fructose + Glucose Beverage: Consumption of a sweet beverage (Fructose:Glucose 1:1, 3g/kg) over 1/2 hour. Blood sampling will occur before and after consumption of beverage.
Period: Overall Study
Arm/Group | Caucasians | South Asians
Started | 19 | 20
Completed | 15 | 15
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 3 | 3
Not completed — screen failure | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Caucasian: Control group: The arm is an oral sugar challenge with blood sampling over 4 hours.
  Fructose + Glucose Beverage: Consumption of a sweet beverage (Fructose:Glucose 1:1, 3g/kg) over 1/2 hour. Blood sampling will occur before and after consumption of beverage.
- South Asians: Experimental group: The arm is an oral sugar challenge with blood sampling over 4 hours.
  Fructose + Glucose Beverage: Consumption of a sweet beverage (Fructose:Glucose 1:1, 3g/kg) over 1/2 hour. Blood sampling will occur before and after consumption of beverage.
- Total: Total of all reporting groups
Arm/Group | Caucasian | South Asians | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (3) | 26 (5) | 27 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Fold Change in Plasma Very Low Density Lipoprotein (VLDL) Triglyceride Palmitate
Description: Fold change in plasma very low density lipoprotein (VLDL) triglyceride palmitate between South Asians and Caucasians from baseline to 4 hours after an oral challenge of fructose:glucose, 1:1.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: fold change
Groups:
- Caucasians: Caucasian control group
- South Asians: South Asian experimental group
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
fold change | 1.24 (0.87) | 1.85 (0.73)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; The equivalence test was used to compare the fold change in plasma VLDL triglyceride palmitate in Caucasians and South Asians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups in the primary outcome- the mean fold change in plasma VLDL triglyceride palmitate, 0-4 hours. A power calculation was based on data obtained in 15 overweight subjects. Assuming a mean absolute difference of 2.7 in South Asians and 1.0 in Caucasians and a standard deviation of 2.0 for both, group sample sizes of 16 and 16 were expected to achieve 80% power to detect a difference of 1.7 using a 2-sided Mann-Whitney test; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 0.61

2. Secondary Outcome: Fold Changes in VLDL Triglycerides in South Asians and Caucasians
Description: 1) A comparison of the fold changes in very low density lipoprotein triglycerides (VLDL TG)in the 2 study groups between 0 and 4 hours.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
fold change | 1.05 (0.56) | 1.44 (0.59)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; The equivalence test was used to compare 1) the fold change in triglycerides in South Asians and Caucasians and 2) the fold change in VLDL triglycerides in South Asians and Caucasians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, t-test, 2 sided

3. Secondary Outcome: Peak Glucose Levels in 2 Study Groups
Description: A comparison of peak levels of glucose at one hour. Glucose is expected to increase after ingestion of glucose/fructose.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
mmol/L | 5.16 (1.83) | 5.61 (1.94)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; The equivalence test is used to compare levels after the sugar beverage of 1) glucose at 1 hour 2) lactate at 1 hour 3) NEFA at 2 hours in South Asians vs Caucasians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Peak Insulin Levels in 2 Study Groups
Description: A comparison of the mean peak insulin level at one hour in each group. Insulin is expected to increase after ingestion of glucose/fructose.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
IU/L | 93 (78) | 111 (45)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, t-test, 2 sided

5. Secondary Outcome: Peak Gastric Inhibitory Protein (GIP) Levels in the 2 Study Groups
Description: A comparison of the mean peak gastric inhibitory protein (GIP) at 2 hours in each group. GIP is expected to increase after ingestion of glucose/fructose.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
ng/L | 277 (90) | 274 (99)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, t-test, 2 sided

6. Secondary Outcome: Correlations Between Fold Change in VLDL TG Palmitate and Other Biomarkers of Carbohydrate and Fat Metabolism
Description: Correlations between fold change in VLDL TG palmitate at 4 hours with other biomarkers of carbohydrate and fat metabolism in each study group.
Time Frame: 4 hours
Measure: Number; unit: r (correlation coefficient)
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
r (correlation coefficient)
  fold change VLDL TG palmitate 4h: VLDL TG 0h | 0.1137 | 0.0127
  fold change VLDL TG palmita 4h:fold change VLDL TG | 0.3339 | 0.3149
  fold change VLDL TG palmitate 4h:total TG 0h | 0.2320 | 0.0359
  fold change VLDL TG palmitat: fold change total TG | 0.3340 | 0.3290
  fold change VLDL TG palmitate 4h:cholesterol 0h | -0.0327 | -0.3910
  fold change VLDL TG palmitat 4h:HDL cholesterol 0h | 0.0883 | -0.3743
  fold change VLDL TG palmita 4h:apolipoprotein B 0h | 0.0587 | -0.1459
  fold change VDLD TG palm 4h:LDL particle number 0h | -0.0045 | -0.0849
  fold change VDLD TG palmitate 4h:LDL size 0h | 0.1508 | 0.0359
  fold change VLDL TG palmitate 4h:glucose 0h | -0.2444 | 0.0188
  fold change VDLD TG palmitate 4h:glucose AUC | 0.2677 | -0.1569
  fold change VDLD TG palmitate 4h:insulin 0h | -0.2778 | -0.1151
  fold change VDLD TG palmitate 4h:insulin AUC | 0.1886 | -0.0070
  fold change VDLD TG palmitate 4h:NEFA 0h | 0.0241 | -0.5689
  fold change VDLD TG palmitate 4h:NEFA nadir 2h | 0.1319 | -0.6151
  fold change VDLD TG palmitate 4h:lactate 0h | 0.1082 | 0.4382
  fold change VDLD TG palmitate 4h:lactate peak 1h | 0.1393 | -0.1953
  fold change VDLD TG palmitate 4h:GIP 0h | -0.3237 | -0.2644
  fold change VDLD TG palmitate 4h:GIP peak 2h | 0.2889 | -0.0453
  fold change VDLD TG palmitate 4h:HOMA-R 0h | -0.2892 | -0.1104
  fold change VDLD TG palmitate 4h:HOMA-B% 0h | -0.2347 | 0.2959
  fold change VDLD TG palmitate 4h:hsCRP 0h | 0.0278 | 0.2463
Statistical Analysis 1: Comparison: Caucasians vs South Asians; The equivalence test was used to analyze the relationship between the primary outcome, fold change in VLDL TG palmitate, and the listed levels of biomarkers of carbohydrate and fat metabolism. The correlation analysis was performed on data from each study group separately; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, Pearson or Spearman's rank test

7. Secondary Outcome: Fold Changes in Triglycerides in 2 Study Groups
Description: 1) A comparison of the fold changes in total triglycerides (TG) in the 2 study groups between 0 and 4 hours.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
fold change | 1.05 (0.56) | 1.43 (0.60)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, t-test, 2 sided

8. Secondary Outcome: Peak Lactate Levels in 2 Study Groups
Description: A comparison of peak levels of lactate (at one hour). Lactate is expected to increase after ingestion of glucose/fructose.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
mmol/L | 3.43 (1.15) | 3.91 (0.75)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, t-test, 2 sided

9. Secondary Outcome: Nadir Non-esterified Fatty Acids (NEFA) Levels in 2 Study Groups
Description: A comparison of the nadir level of non-esterified fatty acids (NEFA at 2 hours). NEFA are expected to decrease.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
mmol/L | 0.09 (0.05) | 0.09 (0.11)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, t-test, 2 sided

10. Secondary Outcome: Peak Glucose in 2 Study Groups
Description: A comparison of peak levels of glucose at 1 hour. Glucose is expected to increase after ingestion of glucose/fructose.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Caucasians | South Asians
Number analyzed (Participants) | 15 | 15
mmol/L | 5.16 (1.83) | 5.61 (1.94)
Statistical Analysis 1: Comparison: Caucasians vs South Asians; Test type: Equivalence — A P value <0.05 was used to determine no equivalence between groups; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 hours per participant.
Arm/Group | Caucasians | South Asians
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caucasians (N=15) | South Asians (N=15)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Mild nausea after ingestion of beverage in one subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes